CLINICAL TRIAL: NCT03591809
Title: The Effect of Combined Exercise Training on Cognitive Functions in Patients With Multiple Sclerosis
Brief Title: Combined Exercise Training in Patients With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Cagla Ozkul, research assistant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 400
Record Dates: First submitted 2018-07-09; First posted 2018-07-19 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Multiple Sclerosis
Keywords: cognitive function; fatigue; quality of life; Functional exercise capacity
MeSH Terms: conditions — Multiple Sclerosis; Fatigue

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, single-blind trial
Who Masked: Outcomes Assessor
Masking Description: To ensure blinding, the assessor physiotherapist will not be aware of the arm to which the subjects belong
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- combined exercise training group (Experimental): The combined exercise training group will be given combined exercise training, consisting of Pilates and aerobic exercise, three times during 8 weeks.
  Interventions: Other: combined exercise training
- Control group (No Intervention): The patients in the control group will not apply an exercise training.

INTERVENTIONS:
Other: combined exercise training — The combined exercise training group will be given combined exercise training, consisting of Pilates and aerobic exercise, three times during 8 weeks.
  Arms: combined exercise training group

SUMMARY:
It is stated that the affected cognitive functions in Multiple Sclerosis are learning, memory, attention, speed of information processing, visuospatial skills, and executive functions. The speed of information processing, visual learning and memory are the most frequently affected components in MS. For this reason, approaches to increase cognitive functions by activating neuroprotective mechanisms such as exercise in patients with MS are needed.

The purpose of this study is to examine the effect of combined exercise training on cognitive functions in patients with MS.

DETAILED DESCRIPTION:
The study was designed as a randomized, controlled, single-blind trial. This study will include patients with MS who 0-5.5 according to the Extended Disability Status Scale (EDSS) and between 18-65 years. The patient will be randomized into a combined training group and a control group. The patients in the control group will not apply an exercise training. The combined exercise training group will be given combined exercise training, consisting of Pilates and aerobic exercise, three times during 8 weeks. Both groups will be reevaluated 8 weeks after the initial assessment.

Statistical analyses will be performed using the SPSS software version 15 (SPSS Inc. Chicago, IL, USA). The pre-training and post-training measurements of groups will be compared with the Wilcoxon Test. The significance level was set at p< 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory
* Stable phase of the disease without relapses in the last 3 month
* EDSS between 2-5,5.

Exclusion Criteria:

* Orthopedic, vision, hearing, or perception problems
* Any cardiovascular or pulmonary disease in which exercise is contraindicated

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2019-10-21 (Actual)

PRIMARY OUTCOMES:
cognitive function | Thirty minutes]
  The Brief Repeatable Battery of Neuropsychological Tests

SECONDARY OUTCOMES:
functional exercise capacity | ten minutes
  The Six-Minute Walking Test (6MWT) was performed to determine functional exercise capacity
Fatigue | five minutes
  Fatigue impact scale will be used to asses fatigue. There are 40 items, each of which is scored 0 (no problem) to 4 (extreme problem), providing a continuous scale of 0-160. It is composed of three subscales that describe how fatigue impacts upon cognitive (10 items), physical (10 items) and psychosocial functioning (10 items). Cognitive functioning concerns concentration, memory, thinking and organization of thoughts. Physical functioning reflects motivation, effort, stamina and coordination. Psychosocial functioning describes the impact of fatigue upon isolation, emotions, workload and coping.A higher score indicates a higher fatigue impact.
Multiple Sclerosis Quality of Life-54 | ten minutes
  The questionnaire consists of 54 questions with 12 sub-sections; physical function, health perceptions, energy/fatigue, role limitations-physical, pain, sexual function, social function, health distress, the overall quality of life, emotional well-being, role limitations-emotional, cognitive function. The summary scores are the physical health composite summary and the mental health composite summary. There is no single overall score for the MSQOL-54. Two summary scores - physical health and mental health - can be derived from a weighted combination of scale scores. In this scale, the scoring of each question is different from each other and a higher score indicates a lower quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Cagla Ozkul, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rao SM, Leo GJ, Bernardin L, Unverzagt F. Cognitive dysfunction in multiple sclerosis. I. Frequency, patterns, and prediction. Neurology. 1991 May;41(5):685-91. doi: 10.1212/wnl.41.5.685. PMID 2027484
- [Background] Rogers JM, Panegyres PK. Cognitive impairment in multiple sclerosis: evidence-based analysis and recommendations. J Clin Neurosci. 2007 Oct;14(10):919-27. doi: 10.1016/j.jocn.2007.02.006. Epub 2007 Jul 30. PMID 17659875
- [Background] Janculjak D, Mubrin Z, Brinar V, Spilich G. Changes of attention and memory in a group of patients with multiple sclerosis. Clin Neurol Neurosurg. 2002 Jul;104(3):221-7. doi: 10.1016/s0303-8467(02)00042-2. No abstract available. PMID 12127658
- [Background] Rosti-Otajarvi EM, Hamalainen PI. Neuropsychological rehabilitation for multiple sclerosis. Cochrane Database Syst Rev. 2014 Feb 11;2014(2):CD009131. doi: 10.1002/14651858.CD009131.pub3. PMID 24515630
- [Background] Cotman CW, Berchtold NC, Christie LA. Exercise builds brain health: key roles of growth factor cascades and inflammation. Trends Neurosci. 2007 Sep;30(9):464-72. doi: 10.1016/j.tins.2007.06.011. Epub 2007 Aug 31. PMID 17765329
- [Background] Smith PJ, Blumenthal JA, Hoffman BM, Cooper H, Strauman TA, Welsh-Bohmer K, Browndyke JN, Sherwood A. Aerobic exercise and neurocognitive performance: a meta-analytic review of randomized controlled trials. Psychosom Med. 2010 Apr;72(3):239-52. doi: 10.1097/PSY.0b013e3181d14633. Epub 2010 Mar 11. PMID 20223924
- [Background] Sangelaji B, Estebsari F, Nabavi SM, Jamshidi E, Morsali D, Dastoorpoor M. The effect of exercise therapy on cognitive functions in multiple sclerosis patients: A pilot study. Med J Islam Repub Iran. 2015 Apr 22;29:205. eCollection 2015. PMID 26157723
- [Background] Romberg A, Virtanen A, Ruutiainen J. Long-term exercise improves functional impairment but not quality of life in multiple sclerosis. J Neurol. 2005 Jul;252(7):839-45. doi: 10.1007/s00415-005-0759-2. Epub 2005 Mar 16. PMID 15765197